CLINICAL TRIAL: NCT02738983
Title: Thoracic Radiotherapy Combined With EGFR-TKI for Wild-type Non-small Cell Lung Cancer
Brief Title: RT Plus EGFR-TKI for Wild-type NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhishuang Zhen, MD, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH04
Record Dates: First submitted 2016-04-04; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer; Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI)
Keywords: Non-small cell lung cancer; epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI); Radiotherapy; wild type
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; icotinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bioradiotherapy (Experimental): Erlotinib (trade name: Tarceva®) (150mg oral daily) or Icotinib (trade name: Conmana®) (125mg oral three times a day) with concurrent radiotherapy to a total radiation dose of 60-66 Gray (Gy).
  Interventions: Drug: Erlotinib (trade name: Tarceva®) or Icotinib (trade name: Conmana®); Radiation: Radiotherapy

INTERVENTIONS:
Drug: Erlotinib (trade name: Tarceva®) or Icotinib (trade name: Conmana®) — Erlotinib (trade name: Tarceva®) (150mg oral daily) or Icotinib (trade name: Conmana®) (125mg oral three times a day).
Radiation: Radiotherapy — Concurrent radiotherapy total dose 60-66 Gy in 2 Gy fractions. One fraction per day, and 5 fractions per week.

SUMMARY:
Concurrent chemoradiotheray is the standard care for patients with locally advanced non-small cell lung cancer (NSCLC), but often accompanying with high toxicity and poor tolerability. Radiosensitization of epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKI) has been proved in preclinical studies, and the safety of TKI combined with thoracic radiotherapy has also been evaluated in several phase II trials. The aim of study is to investigate the efficacy and safety of thoracic radiotherapy combined with TKI in wild-type EGFR patients who refused or unsuitable for concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. NSCLC confirmed by histopathology or cytology;
2. Stage IIA - IV NSCLC ,unresectable and could not tolerate chemoradiotherapy;
3. Has measurable lesion [according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, must have at least one evaluable lesion with the longest dimension >= 10mm; if the evaluable lesion is lymph node, the shortest dimension should be measured and >=15mm];
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
5. Expectancy life >= 3 months;

Exclusion Criteria:

1. Had systemic anit-NSCLC treatments;
2. Had be treated by HER-targeting agents;
3. Had local radiotherapy for NSCLC;
4. Has upper gastrointestinal physiological disorders, or malabsorption syndrome, or intolerance of oral medication, or active peptic ulcer;
5. Diagnosed other malignant tumor besides NSCLC within 5 years prior the study treatment (except having simple surgical resection with 5-year disease free survival, cured in situ of cervical carcinoma, cured basal cell carcinoma and bladder epithelial tumor);
6. Any evidence to indicate moderate or severe chronic obstructive pulmonary disease (COPD);
7. Known hypersensitivity to EGFR-TKI agents or relevant components in the formulation;
8. Uncontrolled eye inflammation or infection, or any potential circumstances lead to eye inflammation or infection;
9. Pregnancy or breast-feeding women;
10. Ingredients mixed with small cell lung cancer patients;
11. Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | week 3-4

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0. | year 0- year 2
  Toxicity of the treatment will be evaluated according to the common toxicity criteria for adverse events version 3.0 (CTCAE v3.0).
Progression-free survival | year 0- year 2
  Progression-free survival (PFS) will be calculated from the date of treatment initiation to the date of documented failure (local recurrence or metastasis occurrence) or the date of the last follow-up for those remaining.
Overall survival | year 0- year 2
  Overall survival (OS) wiil be determined as the time (in months) between the first day of therapy and the last follow-up or the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Shixiu Wu, MD, Study Chair — Hangzhou Cancer Hospital
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided